CLINICAL TRIAL: NCT06970522
Title: Early Detection of Atypical Neuromuscular Development Using Wearable Sensors and Video: A Comparative Analysis of Muscle and Motion
Brief Title: Wearable Sensors to Detect Atypical Muscle Activation in Young Infants
Status: Recruiting | Type: Observational
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Ann & Robert H Lurie Children's Hospital of Chicago (Other); Northwestern University (Other)
Responsible Party: Principal Investigator, Arun Jayaraman, PT, PhD, Principal Investigator, Shirley Ryan AbilityLab
Other Study IDs: 2024 6737
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Neuromuscular Disorders; Motor Development; Muscle Tone
Keywords: Early Detection; Wearable Sensors
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infants with Typical Tone
- Infants with Low Tone

SUMMARY:
The purpose of this study is to see if wearable sensor technology can be used to evaluate muscle activity and/or identify atypical muscle tone in infants up to 48 weeks postmenstrual age (8 weeks corrected age). These sensors are placed on the surface of the skin and record data about a child's body movements and muscle activity.

ELIGIBILITY:
Inclusion Criteria:

* For Infants with low tone:
* Hospitalized in the NICU
* AND >38 weeks post-menstrual age
* AND abnormal normal brain imaging OR Apgar score <7 at five minutes with umbilical cord pH (if obtained) <7.15
* AND 2 or more warning signs for muscle tone or posture using the HNNE short form
* AND legal guardian able and willing to give written consent and comply with study procedures
* For Infants with typical tone:
* Born at 38-41 weeks of gestation
* AND hospitalized after birth in the NICU OR well newborn nursery
* AND infants with appropriate for gestational age birth weight
* AND HNNE exam (short proforma) normal with no warning signs for any parameter
* AND legal guardian able and willing to give written consent and comply with study procedures.

Exclusion Criteria:

* Infants of Both Low Tone and Typical Tone Cohorts:
* Missing or incomplete limbs (such as from amputation or congenital limb defects).
* Open wounds or skin breakdown on the limbs or torso.
* Presence of known genetic syndrome or congenital anomalies requiring surgery or affecting function
* Use of sedative medications (may include phenobarbital if level stable and therapeutic)
* Legal guardian unable to give written consent and comply with study procedures.
* Does not receive medical clearance from a physician to participate in the study if the individual is receiving inpatient care.

Ages: 0 Months to 8 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants presenting with atypical muscle tone based on clinical expertise along with infants expected to have typical development.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Correlation Between EMG Data and Observed Muscle Tone Before 8 Weeks Corrected Age | Before 8 weeks corrected age
  Correlation of EMG sensor data and Hammersmith Neonatal Neurological Exam (HNNE) short form score, assessed before 8 weeks corrected age.

SECONDARY OUTCOMES:
Estimation of Clinical Scores Performed Before 8 Weeks Corrected Age Using EMG Data | Before 8 weeks corrected age
  Error between true clinical test scores and estimated scores using EMG sensor data, assessed before 8 weeks corrected age.

CONTACTS AND LOCATIONS:
Overall Officials: Arun Jayaraman, PT, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (2):
- United States (2):
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Shirley Ryan AbilityLab, Chicago, Illinois